CLINICAL TRIAL: NCT01900678
Title: VLIC-USA: A Single-Center Study of the Safety and Efficacy of the VytronUS Low-Intensity Collimated Ultrasound Ablation System
Brief Title: A Study of the Safety and Efficacy of the VytronUS Low-Intensity Collimated Ultrasound Ablation System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VytronUS, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VLIC-USA; CIV-13-04-010581 (Registry Identifier: EUDAMED)
Record Dates: First submitted 2013-07-09; First posted 2013-07-16 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VytronUS Ablation System (Experimental): Treatment with the VytronUS Ablation System.
  Interventions: Device: VytronUS Ablation System

INTERVENTIONS:
Device: VytronUS Ablation System — Pulmonary vein isolation.

SUMMARY:
The objective of this investigation is to evaluate whether pulmonary vein isolation using the VytronUS ablation system is safe and effective acutely and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years old.
* Recurrent symptomatic paroxysmal atrial fibrillation refractory to at least one antiarrhythmic drug.

Exclusion Criteria:

* Prior pulmonary vein isolation
* Presence of intracardiac thrombus
* Indication of inaccessible pulmonary or cardiac anatomy
* Myocardial infarction, PCI, or cardiac surgery in prior three months
* Moderate to severe valvular disease or prior valve replacement
* NYHA Class IV
* LVEF < 40%
* Previous stroke or TIA
* Serum creatinine > 2.5mg/dL or allergy to intravenous contrast agents
* Existing bleeding diathesis or history of complications with anticoagulation therapy
* Women who are nursing, pregnant, or trying to become pregnant
* Subjects unwilling or unable to provide consent
* Participation in a drug or device trial that would prevent completion of required study procedures
* Active implantable devices
* Major organ system disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Device or procedure related adverse events. | Three months post procedure.

SECONDARY OUTCOMES:
Pulmonary vein isolation. | Three months post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Neuzil, MD, PhD, Principal Investigator — Na Homolce Hospital
Locations (1):
- Na Homolce Hospital, Prague, Czechia